CLINICAL TRIAL: NCT03946631
Title: Immediate Postpartum Screening for Diabetes Mellitus in Women With Gestational Diabetes.
Brief Title: GDM Post Partum Screening
Status: Terminated | Type: Observational
Why Stopped: PI and Practice closed
Sponsor: Pediatrix (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GDM 2019 iris 01-18-0028
Record Dates: First submitted 2019-04-15; First posted 2019-05-10 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Gestational Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fingerstick blood glucose test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Glucose Test - 2hour GTT: Only one arm: intervention group. The intervention is fasting 2 hour glucose tolerance test in the immediate postpartum period. The screening test consists of fingerstick blood glucose testing after a glucose drink. First, a fasting blood glucose finger stick will be performed. Second, the glucose drink is orally ingested containing 75g glucose. The drink is to be orally ingested over 60 seconds. Lastly, fingerstick blood glucose testing is completed at 1 hour post drink and 2 hours post drink.
  Interventions: Diagnostic Test: 2 hour glucose tolerance test using 75g glucose drink

INTERVENTIONS:
Diagnostic Test: 2 hour glucose tolerance test using 75g glucose drink — intervention is a 2 hour glucose tolerance test. Involves oral intake of a 75g glucose drink followed by using point of care testing. Glucose drink is taken after at least 6 hours of fasting. Fingerstick blood glucose testing done at three time points: fasting, one hour post drink and two hours post drink.
  Other Names: fingerstick testing

SUMMARY:
Immediate postpartum screening for diabetes mellitus in women with gestational diabetes

The objective of this study is to determine if screening for type 2 diabetes can be done 24 hours after delivery, versus 6-12 weeks postpartum, in recently delivered women having been diagnosed with gestational diabetes requiring medication therapy in the antecedent pregnancy.

DETAILED DESCRIPTION:
1 Overview The purpose of the project is to determine if screening for diabetes mellitus, in women with gestational diabetes, can be done 24 hours postpartum versus 6-12 weeks postpartum.

Primary Objective: To compare the results from screening for type 2 diabetes 24 hours postpartum versus 6-12 weeks postpartum.

Design and Project Type Prospective cohort study. Women diagnosed with gestational diabetes and receiving anti-hyperglycemic medication therapy will have testing for type 2 DM done 24 hours after delivery. They will also have routine screening for type 2 DM done at 6-12 weeks postpartum.

Description of Intervention The intervention is early screening for type 2 DM which involves oral intake of a 75-- gram (g) glucose drink and subsequent measurement of fasting, 1- hour, and 2- hour postprandial point of care fingerstick s for blood glucose measurement.

Instruments Fingerstick testing will be done with StatStrip Glucose Hospital Meter (Nova Biomedical). This device is used routinely throughout the hospital and has been validated for use in all patients, including the critically ill. Using point of care testing will allow for accurate results with less pain for the patient, as compared to (fingerstick versus venipuncture).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, or recently postpartum, women with the diagnosis of GDM requiring medication therapy after 20 weeks,
* >18 years-old (yo)yo,
* English speaking.

Exclusion Criteria:

* have pre-existing type 2 DM,
* did not require anti-hyperglycemic medication therapy (GDMA1),
* early onset GDM (<20 weeks).
* do not speak English .

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females with current diagnosis of type 2 DM or gestational diabetes
Study Population: Pregnant, or recently postpartum, women with the diagnosis of GDM requiring medication therapy after 20 weeks, >18 years-old (yo), English speaking
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity of early postpartum overt diabetes screening by 2-hour glucose tolerance testing in postpartum women. | 24-48 hours postpartum verses 6-12 weeks postpartum.
  We will compare the sensitivity of a 2-hour oral glucose tolerance test (2HR OGTT) for the detection of overt diabetes when performed within 48 hours of delivery ("early") among postpartum women previously diagnosed with gestational diabetes requiring treatment. The "early" 2HR OGTT result will be compared to the current standard of care of a 2HR OGTT performed at 6-12 weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Wilkes, Study Director — Banner University Medical Center; Kisti Fuller, MD, Principal Investigator — Phoenix Perinatal Associates, Mednax
Locations (1):
- Banner - University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gobl CS, Bozkurt L, Prikoszovich T, Winzer C, Pacini G, Kautzky-Willer A. Early possible risk factors for overt diabetes after gestational diabetes mellitus. Obstet Gynecol. 2011 Jul;118(1):71-78. doi: 10.1097/AOG.0b013e318220e18f. PMID 21691165
- [Background] Su X, Zhang Z, Qu X, Tian Y, Zhang G. Hemoglobin A1c for diagnosis of postpartum abnormal glucose tolerance among women with gestational diabetes mellitus: diagnostic meta-analysis. PLoS One. 2014 Jul 11;9(7):e102144. doi: 10.1371/journal.pone.0102144. eCollection 2014. PMID 25014072
- [Background] Mendez-Figueroa H, Daley J, Breault P, Lopes VV, Paine V, Goldman D, Francis MJ, Delgado B, Coustan DR. Impact of an intensive follow-up program on the postpartum glucose tolerance testing rate. Arch Gynecol Obstet. 2014 Jun;289(6):1177-83. doi: 10.1007/s00404-014-3157-0. Epub 2014 Jan 31. PMID 24481876
- [Background] Kjos SL, Peters RK, Xiang A, Henry OA, Montoro M, Buchanan TA. Predicting future diabetes in Latino women with gestational diabetes. Utility of early postpartum glucose tolerance testing. Diabetes. 1995 May;44(5):586-91. doi: 10.2337/diab.44.5.586. PMID 7729620
- [Background] 5. Biljok VR, Bozicevic S, Lovrencic MV, Car N. Performance of the StatStrip Glucose Meter in Inpatient Management of Diabetes Mellitus. Diabetologia Croatica 2010; 39-3:105-109.
- [Background] Werner EF, Has P, Tarabulsi G, Lee J, Satin A. Early Postpartum Glucose Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2016 Aug;33(10):966-71. doi: 10.1055/s-0036-1583193. Epub 2016 Apr 27. PMID 27120481
- [Background] Dinglas C, Muscat J, Heo H, Islam S, Vintzileos A. Immediate Postpartum Glucose Tolerance Testing in Women with Gestational Diabetes: A Pilot Study. Am J Perinatol. 2017 Oct;34(12):1264-1270. doi: 10.1055/s-0037-1606620. Epub 2017 Sep 14. No abstract available. PMID 28910846
- [Background] Vucic Lovrencic M, Radisic Biljak V, Bozicevic S, Pape-Medvidovic E, Ljubic S. Validation of Point-of-Care Glucose Testing for Diagnosis of Type 2 Diabetes. Int J Endocrinol. 2013;2013:206309. doi: 10.1155/2013/206309. Epub 2013 Dec 8. PMID 24382960